CLINICAL TRIAL: NCT04203511
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of INCMGA00012, an Anti-PD-1 Antibody, in Combination With Chemoradiation in Participants With Unresectable, Stage III Non-Small Cell Lung Cancer (POD1UM-301)
Brief Title: INCMGA00012 in Combination With Chemoradiation in Participants With Stage III Non-Small Cell Lung Cancer (POD1UM-301)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Strategic/Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCMGA 0012-301
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; unresectable; Stage III; PD-1; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; Etoposide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemoradiation therapy + INCMGA00012 (Experimental)
  Interventions: Drug: Retifanlimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Etoposide; Radiation: Radiotherapy
- Chemoradiation therapy + Placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Etoposide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Retifanlimab — INCMGA00012 administered intravenously every 3 weeks on Day 1 of each 21-day cycle for 4 cycles, followed by a consolidation part of INCMGA00012 administered intravenously on Day 1 of each 28-day cycle for up to12 cycles.
  Other Names: INCMGA00012
  Arms: Chemoradiation therapy + INCMGA00012
Drug: Placebo — Placebo administered intravenously every 3 weeks on Day 1 of each 21-day cycle for 4 cycles, followed by a consolidation part of placebo administered intravenously on Day 1 of each 28-day cycle for up to 12 cycles.
  Arms: Chemoradiation therapy + Placebo
Drug: Pemetrexed — Pemetrexed administered intravenously every 3 weeks on Day 1 of each cycle with either carboplatin or cisplatin (nonsquamous NSCLC only) for 2 cycles (if radiation therapy is started on Cycle 1 Day 1) or 3 cycles (if radiation therapy is started after Cycle 1).
Drug: Cisplatin — Cisplatin administered intravenously every 3 weeks on Day 1 of each cycle with either etoposide or pemetrexed (nonsquamous NSCLC only) for 2 cycles (if radiation therapy is started on Cycle 1 Day 1) or 3 cycles (if radiation therapy is started after Cycle 1).
Drug: Carboplatin — Carboplatin administered intravenously every 3 weeks on Day 1 of each cycle with either pemetrexed (nonsquamous NSCLC only) or paclitaxel for 2 cycles (if radiation therapy is started on Cycle 1 Day 1) or 3 cycles (if radiation therapy is started after Cycle 1).
Drug: Paclitaxel — Paclitaxel administered intravenously every 3 weeks on Days 1, 8, and 15 of each cycle with carboplatin for 2 cycles (if radiation therapy is started on Cycle 1 Day 1) or 3 cycles (if radiation therapy is started after Cycle 1).
Drug: Etoposide — Etoposide administered intravenously every 3 weeks on Days 1-3 of each cycle with cisplatin for 2 cycles (if radiation therapy is started on Cycle 1 Day 1) or 3 cycles (if radiation therapy is started after Cycle 1).
Radiation: Radiotherapy — Total dose of 60 Gy ± 10% (54 to 66 Gy) in 2 Gy daily fractions.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of INCMGA00012 in combination with chemoradiation therapy (CRT) in participants with unresectable, Stage III non-small cell lung cancer (NSCLC). The study will randomize approximately 360 participants in a 2:1 ratio into the INCMGA00012 in combination with CRT followed by consolidation therapy with INCMGA00012 treatment group and placebo in combination with CRT followed by consolidation therapy with placebo treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC that is locally advanced and unresectable.
* Adequate tumor sample from fresh biopsy or archival tissue block must be available.
* Evaluable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Receipt of cancer treatment for this malignancy, including but not limited to radiation therapy, investigational agents, chemotherapy, and immunotherapy for disease under consideration.
* Recent major surgery within 4 weeks before entry into the study.
* Any medical contraindication to platinum-based doublet chemotherapy.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic consolidation doses of corticosteroids (> 10 mg/day of prednisone or equivalent).
* Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Mixed small cell and NSCLC histology.
* Evidence of interstitial lung disease or active noninfectious pneumonitis.
* Participants who are HIV-positive.
* History of organ transplant, including allogeneic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-31 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 3 years.
  Defined as the time from randomization until disease progression, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as determined by blinded independent central review (BICR), or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 3 years.
  Defined as the time from randomization until death due to any cause.
Objective response rate (ORR) | Up to approximately 3 years.
  Defined as the percentage of participants having a complete response or partial response per RECIST v1.1 based on BICR.
Duration of response (DOR) | Up to approximately 3 years.
  Defined as the time from the first documented response (complete response or partial response) according to RECIST v1.1 until disease progression or death due to any cause.
Number of treatment-emergent adverse events | Up to approximately 3 years.
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study treatment.
Cmax of INCMGA00012. | Cycle 1 Day 1, Cycle 2 Day 1 and Consolidation Cycle 1 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, and Cycle 12 Day 1, up to approximately 18 months.
  Maximum observed plasma or serum concentration.
tmax of INCMGA00012. | Cycle 1 Day 1, Cycle 2 Day 1 and Consolidation Cycle 1 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, and Cycle 12 Day 1, up to approximately 18 months.
  Time to maximum concentration.
Cmin of INCMGA00012. | Cycle 1 Day 1, Cycle 2 Day 1 and Consolidation Cycle 1 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, and Cycle 12 Day 1, up to approximately 18 months.
  Minimum observed plasma or serum concentration over the dose interval.
AUC0-t of INCMGA00012. | Cycle 1 Day 1, Cycle 2 Day 1 and Consolidation Cycle 1 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, and Cycle 12 Day 1, up to approximately 18 months.
  Area under the plasma or serum concentration curve.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation

IPD SHARING:
Plan to Share IPD: No